CLINICAL TRIAL: NCT04925167
Title: Safety and Efficacy of Argatroban Applicated in Anticoagulation of V-V ECMO: A Randomized Controlled Study
Brief Title: Safety and Efficacy of Argatroban Applicated in Anticoagulation of V-V ECMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Bing Sun, Professor, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Argatroban in V-V ECMO
Record Dates: First submitted 2021-06-11; First posted 2021-06-14 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — argatroban; Heparin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- argatroban group (Experimental): Patients received argatroban for anticoagulation during V-V ECMO.
  Interventions: Drug: Argatroban
- UFH group (Active Comparator): Patients received UFH for anticoagulation during V-V ECMO.
  Interventions: Drug: unfractionated heparin

INTERVENTIONS:
Drug: Argatroban — Argatroban continuous intravenous injection maintained APTT at 1.5 times of baseline.
  Other Names: Novastan
  Arms: argatroban group
Drug: unfractionated heparin — unfractionated heparin continuous intravenous injection maintained APTT at 1.5 times of baseline.
  Arms: UFH group

SUMMARY:
Unfractionated heparin is most common in the anticoagulation management of V-V ECMO. However, many side effects of unfractionated heparin, such as HIT, antithrombin deficiency, etc seriously affects the prognosis of patients. Argatroban is kind of direct thrombin inhibitors, which could be used used as an alternative anticoagulant of unfractionated heparin when HIT or antithrombin deficiency, etc. At present, there is no power enough evidence for the application of argatroban in V-V ECMO. This study aims to evaluat the safety and effectiveness of argatroban in the anticoagulation management of V-V ECMO compared with unfractionated heparin.

ELIGIBILITY:
Inclusion Criteria:

* age older than 18 years old; received V-V ECMO because of sevever respiratory failure

Exclusion Criteria:

* anticoagulant contraindications; Confirmed or suspected, or previously diagnosed with heparin induced thrombocytopenia; Cerebral infarction or suspected patients; Patients with severe liver dysfunction; Allergic to heparin or argatroban; hemophilia; Unwilling or unable to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
incidence of ECMO related thrombotic events | 14 days
  the incidence of ECMO related thrombotic events, such as membrane oxygenator or tube thrombosis.

CONTACTS AND LOCATIONS:
Overall Officials: Bing Sun, MD, Principal Investigator — Beijing Chao Yang Hospital
Locations (1):
- Bing Sun, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Study protocal, statistical analysis plan, informed consent form and clinical study report will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1 year after the study completed.
Access Criteria: Contact PI by email with reasonable reasons.